CLINICAL TRIAL: NCT03344003
Title: Immune Tolerance Induction in Haemophilia A Patients Using Wilate or Nuwiq - A Canadian Study
Brief Title: Immune Tolerance Induction in Haemophilia A Patients Using Wilate or Nuwiq
Acronym: PREVAIL
Status: Terminated | Type: Observational
Why Stopped: Study terminated as enrolled patients rolled over into a large international study in the same indication
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: WIL-26
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — von Willebrand Factor; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wilate or Nuwiq prospective cohort: Evaluable haemophilia A patients with an inhibitor against FVIII enrolled prospectively
  Interventions: Drug: Wilate or Nuwiq
- Wilate or Nuwiq retrospective cohort: Evaluable haemophilia A patients with an inhibitor against FVIII enrolled retrospectively
  Interventions: Drug: Wilate or Nuwiq

INTERVENTIONS:
Drug: Wilate or Nuwiq — Wilate or Nuwiq administered via intravenous injection
  Other Names: Wilate: Human von Willebrand factor / human coagulation factor VIII. Nuwiq: recombinant factor VIII (rhFVIII)

SUMMARY:
Uncontrolled, multi-centre, non-interventional study with a prospective and a retrospective cohort, to evaluate the efficacy of Wilate or Nuwiq in achieving complete or partial immune tolerance induction (ITI) success in severe and moderate haemophilia A patients with inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Male patients of any age with moderate or severe haemophilia A.
* Patients with a first occurrence of inhibitors, inhibitors refractory to previous ITI attempt(s), or relapsed inhibitors to FVIII, with an inhibitor titre of ≥0.6 BU measured on 2 separate occasions at least 2 weeks apart.
* Informed written consent from the patient and/or the patient's parent(s) or legal guardian(s)

For patients in the prospective cohort:

* Patients who are currently on Wilate or Nuwiq ITI, have just initiated ITI, or are planned to initiate ITI treatment with Wilate or Nuwiq.

For patients in the retrospective cohort:

* Patients having received Wilate or Nuwiq ITI before entry into this study. Retrospective data will be collected for a maximum of 3 years before enrolment into the study. To be eligible, the following information is needed:
* Wilate or Nuwiq treatment details (start date, dose, treatment frequency, and dose change).
* Reliably documented bleeding frequency.
* FVIII inhibitor titres.
* FVIII half-life.
* FVIII IVR.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

* Congenital or acquired bleeding disorders other than haemophilia A.
* A history of hypersensitivity to blood products and/or plasma-derived FVIII concentrates.
* Inability to speak/read English or French well enough to provide consent and adhere to the study.
* People who are receiving other non-factor therapies, e.g. concizumab

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of at least 80 patients were planned, at least 40 in the prospective cohort and 40 in the retrospective cohort. Due to study termination, only 14 patients were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sri Adapa, Study Director — Octapharma
Locations (3):
- Canada (3):
  - Stollery children's hospital, University of Alberta, Edmonton, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hamilton Health Science center, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wilate® Retrospective Cohort: The retrospective cohort was made up of 8 patients who had received Wilate immune tolerance induction (ITI) therapy within 3 years of enrolment. All patients had evaluable hemophilia A with an inhibitor against FVIII. The treatment regimen, doses, dosing intervals and dose adjustments were determined at the discretion of the treating physician. A usual dose for long-term prophylaxis against bleeding in patients with severe hemophilia A is 20 to 40 IU of factor VIII per kg body weight at intervals of 2 to 3 days.
  All enrolled patients were treated with Wilate. No patient discontinued the study before the study was terminated.
- Wilate® Prospective Cohort: The prospective cohort was made up of 6 patients who were currently receiving Wilate ITI, had just initiated ITI, or were planned to initiate ITI treatment with Wilate. All patients had evaluable hemophilia A with an inhibitor against FVIII. The treatment regimen, doses, dosing intervals and dose adjustments were determined at the discretion of the treating physician. A usual dose for long-term prophylaxis against bleeding in patients with severe hemophilia A is 20 to 40 IU of factor VIII per kg body weight at intervals of 2 to 3 days.
  All enrolled patients were treated with Wilate. No patient discontinued the study before the study was terminated.
Period: Overall Study
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Started | 8 | 6
Completed (Study terminated prior to planned completion) | 6 | 6
Not Completed | 2 | 0
Not completed — Switched to alternative treatment | 1 | 0
Not completed — Experienced a better response with recombinant activated factor VII (rFVIIa) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Wilate® Retrospective Cohort: The population consists of all patients who had received Wilate immune tolerance induction (ITI) therapy within 3 years of enrolment.
- Wilate® Prospective Cohort: The population consists of all patients who were currently on Wilate ITI, had just initiated ITI, or were planned to initiate ITI treatment with Wilate.
- Total: Total of all reporting groups
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (5.2) | 14.8 (7.3) | 12.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 5 | 4 | 9
  Other | 1 | 2 | 3
  Missing | 1 | 0 | 1
Blood type [Count of Participants; unit: Participants]
  O | 3 | 2 | 5
  A | 2 | 2 | 4
  B | 1 | 0 | 1
  AB | 1 | 2 | 3
  Missing | 1 | 0 | 1
Severity of hemophilia A [Count of Participants; unit: Participants] — Moderate Hemophilia was defined as the patient having a FVIII activity level of between 1-5%. Severe Hemophilia was defined as the patient having a FVIII activity level below 1%.
  Participants
    Mild | 5 | 2 | 7
    Moderate | 1 | 1 | 2
    Severe | 1 | 3 | 4
    Missing | 1 | 0 | 1
FVIII mutation [Count of Participants; unit: Participants]
  Intron 22 Inversion | 3 | 3 | 6
  Intron 1 Inversion | 1 | 0 | 1
  Missense mutations | 0 | 1 | 1
  Unknown | 3 | 2 | 5
  Missing | 1 | 0 | 1
Previous inhibitor treatment [Count of Participants; unit: Participants]
  Yes | 6 | 4 | 10
  No | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Moderate and Severe Haemophilia A Patients With Inhibitors Achieving Complete or Partial Immune Tolerance Induction (ITI) Success
Description: ITI success will be determined using predefined success criteria to analyze the proportion of patients achieving complete or partial ITI success. Complete success is defined by achieving all of the following variables: 1) Inhibitor titre <0.6BU (at least 2 separate blood samplings) assessed using the modified Bethesda assay; 2) Incremental in vivo recovery (IVR) of FVIII in the normal range (≥66% of normal); 3) FVIII half-life ≥6 hours Wilate infusion. Partial success is defined as two of the three criteria being met, whilst partial response is defined as one of the three criteria being met. Partial failure is defined as none of the three criteria are met, but the inhibitor titre has decreased to <5 BU; complete failure is defined as none of the three criteria are met, and the inhibitor titre is still ≥5 BU.
Time Frame: From ITI start until termination of study, a maximum of 2 years
Population: Due to study termination, efficacy data was not collected for enrolled patients in the prospective cohort
Measure: Count of Participants; unit: Participants
Groups:
- Wilate® Respective Cohort: This cohort was made up of patients who had received Wilate immune tolerance induction (ITI) therapy within three years of enrolment
- Wilate® Prospective Cohort: This cohort consisted of patients who were currently on Wilate ITI, had just initiated ITI, or were planned to initiate ITI treatment with Wilate
Arm/Group | Wilate® Respective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 8 | 0
Participants
  Complete success | 7 | 0
  Partial success | 0 | 0
  Partial failure | 0 | 0
  Complete failure | 1 | 0

2. Secondary Outcome: Time Necessary to Achieve Complete or Partial ITI Success
Description: Time to achieve complete or partial ITI success will be determined using predefined success criteria. Complete success is defined by achieving all of the following variables: 1) Inhibitor titre <0.6 BU (at least 2 separate blood samplings) assessed using the modified Bethesda assay; 2) Incremental IVR of FVIII in the normal range (≥66% of normal) ; 3) FVIII half-life ≥6 hours. Wilate infusion. Partial success is defined as two of the three criteria being met, whilst partial response is defined as one of the three criteria being met. Partial failure is defined as none of the three criteria are met, but the inhibitor titre has decreased to <5 BU; complete failure is defined as none of the three criteria are met, and the inhibitor titre is still ≥5 BU.
  0 participants analysed for this outcome due to termination of study.
Time Frame: A maximum period of 5 years from ITI start
Population: Due to study termination, data was not collected for enrolled patients in either cohort. Therefore, 0 participants were analysed for this outcome
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: In Case of Complete or Partial ITI Success, Duration of Immune Tolerance
Description: Time from start of ITI success to end of study period
Time Frame: A maximum period of 5 years from ITI start
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Bleeding Frequency While on Wilate or Nuwiq ITI Treatment
Description: Bleeding episodes occurring during the study period will be documented by the patient or their parents in a patient study diary.
Time Frame: A maximum period of 5 years from ITI start
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Association of Inhibitor Titres With the Probability of ITI Success
Description: Inhibitor titre will be assessed at the start of and throughout ITI treatment, including peak inhibitor titres, with the probability of ITI success.
  ITI success will be determined using predefined success criteria. Complete success is defined by achieving all of the following variables: 1) Inhibitor titre <0.6 BU (at least 2 separate blood samplings) assessed using the modified Bethesda assay; 2) Incremental IVR of FVIII in the normal range (≥66% of normal) ; 3) FVIII half-life ≥6 hours. Wilate or Nuwiq infusion. Partial success is defined as two of the three criteria being met, whilst partial response is defined as one of the three criteria being met. Partial failure is defined as none of the three criteria are met, but the inhibitor titre has decreased to <5 BU; complete failure is defined as none of the three criteria are met, and the inhibitor titre is still ≥5 BU.
Time Frame: A maximum period of 5 years from ITI start
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Use of Bypassing Agents Before and During ITI Treatment With Wilate or Nuwiq
Description: Use of bypassing agents is at the discretion of the Investigator, either to treat bleeding or to provide prophylactic therapy. As long as the patient's inhibitor level is ≥0.6 Bethesda units (BU), treatment of BEs may, in addition to FVIII treatment, require the administration of activated prothrombin complex concentrates (aPCC) or recombinant FVIIa.
Time Frame: 12 months before the start of ITI with Wilate or Nuwiq to a maximum of 5 years from starting ITI with Wilate or Nuwiq
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Use of Emicizumab (Hemlibra) During ITI Treatment With Wilate or Nuwiq
Description: The dosing and frequency of emicizumab (Hemlibra) used is at the discretion of the Investigator. As a general guidance, the recommended dose is 3mg/kg once weekly for the first 4 weeks, followed by 1.5mg/kg once weekly, administered as a subcutaneous injection, as per the product monograph.
Time Frame: A maximum period of 5 years from ITI start
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Relapse Rate Following Complete or Partial Successful ITI Using Wilate or Nuwiq
Description: Reoccurrence of >0.6 BU in at least 2 consecutive blood samples after having reached the prophylactic treatment phase; a further ITI initiation (re-start) with Wilate or Nuwiq is at the discretion of the Investigator.
Time Frame: A maximum period of 5 years from ITI start
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Relapse Following Complete or Partial Successful ITI Using Wilate or Nuwiq
Description: Time to reoccurrence of >0.6 BU in at least 2 consecutive blood samples after having reached the prophylactic treatment phase; a further ITI initiation (re-start) with Wilate or Nuwiq is at the discretion of the Investigator.
Time Frame: A maximum period of 5 years from ITI start
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Adherence With the ITI Regimen
Description: During ITI, any injections of Wilate or Nuwiq will be recorded in the patient study diary. The treating physician will review and verify the information provided by the patient.
Time Frame: A maximum period of 5 years from ITI start
Population: as for outcome 2
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse drug reactions were monitored throughout the study from first treatment through to study termination, a maximum of 2 years
Description: There were no treatment-related ADRs during the study
Arm/Group | Wilate® Retrospective Cohort | Wilate® Prospective Cohort
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/6
Other Adverse Events (participants affected / at risk) | 0/8 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wilate® Retrospective Cohort (N=8) | Wilate® Prospective Cohort (N=6)
Device-related infection (Infections and infestations) | 1 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wilate® Retrospective Cohort (N=8) | Wilate® Prospective Cohort (N=6)
Pyrexia (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03344003/Prot_SAP_000.pdf